CLINICAL TRIAL: NCT05695391
Title: A Phase 3 Study of the Safety and Efficacy of Coagulation Factor VIIa (Recombinant) for the Prevention of Excessive Bleeding in Patients With Congenital Hemophilia A or B With Inhibitors to Factor VIII or IX Undergoing Elective Major Surgical Procedures
Brief Title: A Phase 3 Study of the Safety and Efficacy of Coagulation Factor VIIa (Recombinant) for the Prevention of Excessive Bleeding in Patients With Congenital Hemophilia A or B With Inhibitors to Factor VIII or IX Undergoing Elective Major Surgical Procedures SCOPE HIM
Acronym: SCOPE HIM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Feasibility considerations - extended timelines to complete recruitment
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F7TG2202
Record Dates: First submitted 2022-12-21; First posted 2023-01-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Factor VII

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Coagulation Factor VIIa (Recombinant) (Experimental)
  Interventions: Biological: Coagulation Factor VIIa (Recombinant)

INTERVENTIONS:
Biological: Coagulation Factor VIIa (Recombinant) — LR769

SUMMARY:
This is an interventional, prospective, international, multicenter, single-arm, Phase 3, and sequential efficacy and safety study in adolescents and adults with congenital hemophilia A or B with inhibitors to factor VIII (FVIII) or factor IX (FIX) undergoing elective major surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study:

1. be male with a diagnosis of congenital hemophilia A or B of any severity
2. have one of the following:

   1. current positive inhibitor test BU ≥5 (as confirmed at screening by the institutional lab) or history of high-responding inhibitors (BU ≥5) not further successfully treated by Immune Tolerance Induction OR
   2. a condition precluding the use of FVIII or FIX products to treat or prevent bleeding such as a previous anamnestic response after exposure to factor concentrates or a previous failure to respond to FVIII or FIX concentrates
3. be ≥12 years to ≤65 years of age on the day of informed consent
4. be scheduled for an elective major surgical procedure as defined in the study protocol (see Table ''Definitions for the specific purpose of Study F7TG2202'')
5. have Hb ≥ 12 g/dL
6. be capable of understanding and willing to comply with the conditions of the protocol OR in the case of a patient under the age of legal majority, parent(s)/legal guardian(s) must be capable of understanding and willing to comply with the conditions of the protocol
7. have read, understood, and provided written informed consent (patient or parent(s)/legal guardian(s) if the patient is minor according to local regulation) and, where applicable according to local regulation, patient's assent if the patient is minor -

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. have any coagulation disorder other than hemophilia A or B
2. be immunosuppressed (i.e. the patient should not be receiving systemic immunosuppressive medication; CD4+ cell counts at screening should be >200/μL)
3. known intolerance to LR769 or any of its excipients
4. currently receiving immune tolerance induction (ITI) therapy
5. have a known or suspected allergy or hypersensitivity to rabbits or rabbit proteins
6. have platelet count <100,000/μL
7. have received an investigational drug within 30 days or within 5 half-lives of that investigational drug, whichever is longer, of the planned first LR769 administration, or be expected to receive such drug during participation in this study. Patients who have received fitusiran in a clinical study may not participate in this clinical study for 6 months since the last dose and if they have an antithrombin III level not in the normal range at screening.
8. for patients using emicizumab, have received during the last 6 months or currently receiving a maintenance dosing regimen of emicizumab different from the indicated one ± 10% of approved dose), i.e. different from 1.5 mg/kg once weekly (±10%), 3 mg/kg (±10%) every two weeks or 6 mg/kg (±10%) every four weeks
9. for patients using emicizumab, currently be any plans, or notes in the patient's medical records that would suggest the need to increase or decrease emicizumab dosing due to antidrug antibodies (ADAs), reduced PK, or coagulation/safety-related issues (e.g. lack of response, or potential/actual thromboembolic concerns, etc)
10. have a clinically relevant hepatic (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] >3 times the upper limit of normal [ULN]) and/or renal impairment (creatinine >2 times the ULN)
11. have a history of arterial and/or venous thromboembolic events (such as myocardial infarction, ischemic strokes, transient ischemic attacks, DVT, or PE) within 2 years prior to the planned first dose of LR769, uncontrolled arrhythmia, or current New York Heart Association (NYHA) functional classification score of stages II - IV
12. have an active malignancy (those with non-melanoma skin cancer are allowed)
13. have any life-threatening disease or other disease or condition which, according to the investigator's judgment, could imply a potential hazard to the patient, or interfere with the study participation or study outcome (e.g. chronic, unmanaged hepatitis infection)
14. be using aspirin, non-steroidal anti-inflammatory drugs (NSAIDS), herbs, natural medications, or other drugs with platelet inhibitory properties within one week prior to surgery and for the duration of treatment with LR769
15. have active gastric or duodenal ulcer disease
16. have received a FVII- or FVIIa-containing product (either plasma derived or recombinant) within 24 hours prior to administration of LR769
17. have a contraindication to antifibrinolytics
18. have planned combined major surgeries at the same time or have already been enrolled and treated for a previous elective major surgery in the same SCOPE HIM study
19. be administered pharmacologic thromboprophylaxis within 5 half-lives of that medication before surgery or for the duration of treatment with LR769 -

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
proportion of successfully at wound closure | at wound closure
  proportion of successfully treated major procedures defined by a good or excellent global hemostatic response.
proportion of successfully at 24 hours after surgery | at 24 hours after surgical wound closure
  proportion of successfully treated major procedures defined by a good or excellent global hemostatic response.
proportion of successfully at 120 hours after surgery | at 120 hours after surgical wound closure
  proportion of successfully treated major procedures defined by a good or excellent global hemostatic response.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel ESCOBAR, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (15):
- United States (5):
  - Orthopaedic Institute for Children - Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Tulane Univertsity School of Medecine, New Orleans, Louisiana
  - M Health Fairview Center for bleeding and Clotting disorders, Minneapolis, Minnesota
  - University of Texas Health Science Center at Houston, Houston, Texas
- Malaysia (2):
  - Hospital Queen Elisabeth - Kota Kinabalu, Kota Kinabalu, Sabah Province
  - Hospital Ampang, Ampang, Selangor Province
- Hospital Universitario Dr. José Eleuterio González de Nuevo León, Monterrey, Nuevo León, Mexico
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa
- Thailand (2):
  - Chiang Mai University, Chiang Mai
  - Maharaj Nakorn Chiangmai Hospital, Chiangmai University, Chiang Mai
- Turkey (Türkiye) (4):
  - Acibadem Adana Hospital, Seyhan, Adana
  - Hacettepe Üniversitesi Rektörlüğü Sihhiye, Altındağ, Ankara
  - Istanbul Üniversitesi Onkoloji Enstitusu, Fatih, Istanbul
  - Karadeniz Teknik Üniversitesi, Trabzon, Trabzon